CLINICAL TRIAL: NCT02742012
Title: A Multicenter Validation Study of a Multimodal Indicator of Anesthesia Calculated From the Electroencephalogram and Standard Monitoring Parameters
Brief Title: Validation of a Multimodal Indicator of Depth of Anesthesia
Status: Completed | Type: Observational
Sponsor: Technical University of Munich (Other)
Responsible Party: Principal Investigator, Andreas Ranft, Dr. med., Technical University of Munich
Other Study IDs: AMI-1250-KIE-0250-I
Record Dates: First submitted 2015-06-25; First posted 2016-04-18 (Estimated); Last update posted 2018-09-11 (Actual); Status verified 2018-09

CONDITIONS: Anesthesia
Keywords: electroencephalogram; hemodynamic monitoring; respiratory monitoring

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: the study is observational — the study is observational

SUMMARY:
The present study is designed to validate an multimodal indicator of anesthetic depth (Schneider G et al. 2014, Anesthesiology 120, 819-28).

The indicator previously developed shall now be tested on an independent set of data.

The investigators will include 250 patients undergoing general anesthesia in 3 German tertiary care centers.

The design is strictly observational - the anesthetic regime is at the discretion of the clinician and will not be influenced.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years
* elective surgery under general anesthesia
* anticipated operating time of about one hour or longer
* ASA physical status I-III
* written informed consent

Exclusion Criteria:

* chronic intake of CNS affecting drugs
* alcohol or drug abuse in the last three months
* CNS or psychiatric disease
* hardness of hearing or deafness
* abnormal gastrointestinal motility
* non-adherence to fasting guidelines, emergency surgery
* anticipated difficult airway
* pregnancy
* cardiac surgery and surgery involving the head and/or neck
* postoperatively prolonged intubation
* pre- and/or postoperative intensive care treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 250 adult patients scheduled for elective surgery under general anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 257 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
ability of the multimodal indicator of anesthetic depth to discriminate between consciousness and unconsciousness | 1 minute

SECONDARY OUTCOMES:
the indicator's ability to discriminate between consciousness, surgical anesthesia and deep anesthesia | 1 minute

CONTACTS AND LOCATIONS:
Overall Officials: Eberhard F Kochs, MD, Study Chair — Klinikum rechts der Isar Technische Universität München
Locations (3):
- Germany (3):
  - Klinik für Anästhesiologie, Bonn
  - Klinikum rechts der Isar, Department of Anesthesiology, Munich
  - Klinik für Anästhesiologie am Helios Klinikum, Wuppertal